CLINICAL TRIAL: NCT04846920
Title: A Phase 1, Dose-escalation Study to Evaluate Safety and Tolerability of Belzutifan (MK-6482) in Participants With Advanced Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: A Study of Belzutifan (MK-6482) in Participants With Advanced Clear Cell Renal Cell Carcinoma (MK-6482-018)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 6482-018; MK-6482-018 (Other: MSD)
Record Dates: First submitted 2021-04-07; First posted 2021-04-15 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Hypoxia inducible factor (HIF); Hypoxia inducible factor 2 alpha (HIF-2α)
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — belzutifan

STUDY DESIGN:
Intervention Model Description: The "Belzutifan 160 mg BID", "Belzutifan 160 mg TID" and "Belzutifan 200 mg TID" study arms will be enrolled sequentially; the "Belzutifan 120 mg QD" study arm will be enrolled in parallel to the "Belzutifan 160 mg BID", "Belzutifan 160 mg TID" and "Belzutifan 200 mg TID" arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Belzutifan 160 mg BID (Experimental): Participants will receive belzutifan 160 mg orally twice daily (BID). Treatment will continue until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan
- Belzutifan 160 mg TID (Experimental): Participants will receive belzutifan 160 mg orally three times daily (TID). Treatment will continue until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan
- Belzutifan 200 mg TID (Experimental): Participants will receive belzutifan 200 mg orally TID. Treatment will continue until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan
- Belzutifan 120 mg QD (Experimental): Participants will receive belzutifan 120 mg orally once daily (QD). Treatment will continue until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — 40 mg tablet administered orally at a dose of 160 mg, 200 mg, or 120 mg.
  Other Names: MK-6482; PT2977; WELIREG™

SUMMARY:
The goal of this study is to evaluate the safety, tolerability and pharmacokinetics of escalating doses of belzutifan as second line positive (2L+) treatment in participants with advanced clear cell renal cell carcinoma (ccRCC).

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically-confirmed diagnosis of unresectable, locally advanced/metastatic RCC with clear cell component (with or without sarcomatoid features) (may include participants with a diagnosis of von Hippel-Lindau [VHL] associated ccRCC).
* Has experienced disease progression on or after having received at least one previous systemic treatment for advanced ccRCC.
* Shows adequate organ function.
* Male participants are eligible to participate if they are abstinent from heterosexual intercourse or agree to use contraception during the intervention period and for at least 7 days after the last dose of study intervention.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and is not a woman of childbearing potential (WOCBP) or is a WOCBP and using contraception or is abstinent from heterosexual intercourse during the intervention period and for at least 30 days after the last dose of study intervention.

Exclusion Criteria:

* Has hypoxia, or requires intermittent supplemental oxygen, or requires chronic supplemental oxygen.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in situ cancers.
* Has any history of or current brain or meningeal metastasis.
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass graft surgery (CABG) ≤6 months from Day 1 of study drug administration, or New York Heart Association Class III or IV congestive heart failure. Medically controlled arrhythmia stable on medication is permitted.
* Has moderate to severe hepatic impairment.
* Has an active infection requiring therapy (includes tuberculosis).
* Has known human immunodeficiency virus (HIV) and/or hepatitis B or C infections or is known to be positive for hepatitis B surface antigen (HBsAg)/hepatitis B virus (HBV) deoxy ribonucleic acid (DNA) or hepatitis C antibody or ribonucleic acid (RNA).
* Has a history or current evidence of a gastrointestinal (GI) condition (eg, inflammatory bowel disease, Crohn's disease, ulcerative colitis) or impaired liver function.
* Has had major surgery ≤3 weeks prior to first dose of study intervention.
* Has received prior treatment with belzutifan.
* Has received any type of systemic anticancer antibody (including investigational antibody) ≤4 weeks prior to the first dose of study intervention.
* Has recovered from all AEs due to previous therapies to ≤ Grade 1 or baseline. Participants with a ≤ Grade 2 neuropathy may be eligible.
* Has received prior radiotherapy within 2 weeks prior to randomization.
* Has received colony-stimulating factors (CSFs) (e.g., granulocyte-CSF [G-CSF], granulocyte monocyte-CSF [GM-CSF] or recombinant erythropoietin [EPO]) ≤28 days prior to the first dose of study intervention.
* Has participated and received study intervention in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been at least 4 weeks since the last dose of the previous investigational agent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2026-07-21 (Estimated); Study Completion 2026-07-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Experience at Least One Adverse Event (AE) | Up to ~49.5 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported.
Percentage of Participants Who Discontinue Study Treatment Due to an AE | Up to ~48.5 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study treatment due to an AE will be reported.
Percentage of Participants Who Modify or Interrupt Study Treatment Due to an AE | Up to ~48.5 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who modify or interrupt study treatment due to an AE will be reported.
Percentage of Participants Who Experience at Least One Dose-limiting Toxicity (DLT) | Up to ~21 days
  A DLT consists of one or more of the following toxicities: (1) Grade 3 or 4 hypoxia or dyspnea (2) Grade 3 or 4 nausea, vomiting, or diarrhea if persistent for >48 hours despite therapy (3) Grade 3 or 4 cardiovascular, vascular, or thrombotic events (4) Nonhematologic AE ≥Grade 3 in severity (5) Grade 4 nonhematologic toxicity (6) Grade 3 or 4 hematologic toxicities (7) Grade 3 or 4 febrile neutropenia (8) Grade 3 or 4 nonhematologic laboratory value (9) >2 weeks delay in dosing due to intervention-related toxicity (10) Intervention-related toxicity causing intervention discontinuation in the first 21 days of dosing (11) Missing >20% of belzutifan doses due to drug-related AEs in the first 21 days. (12) Grade 5 toxicity. The percentage of participants who experience at least one DLT will be reported.

SECONDARY OUTCOMES:
Area Under the Plasma Concentration Time Curve (AUC) of Belzutifan | Day 1, Day 21: pre-dose, 0.5, 1, 1.5, 2, 4, and 6 hours post-dose; Day 2: pre-dose and 2 hours post-dose
  AUC is a measure of plasma drug concentration and time and is estimated as the area under the plot of plasma concentration against time after belzutifan administration. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine AUC.
Maximum Observed Plasma Concentration (Cmax) of Belzutifan | Day 1, Day 21: pre-dose, 0.5, 1, 1.5, 2, 4, and 6 hours post-dose; Day 2: pre-dose and 2 hours post-dose
  Cmax is the maximum concentration of belzutifan observed in plasma. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmax.
Minimum Observed Plasma Concentration (Cmin) of Belzutifan | Day 1, Day 21: pre-dose, 0.5, 1, 1.5, 2, 4, and 6 hours post-dose; Day 2: pre-dose and 2 hours post-dose
  Cmin is the minimum concentration of belzutifan observed in plasma after its administration and just prior to administration of a subsequent dose. Blood samples collected pre dose and at multiple timepoints post dose will be used to determine Cmin.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center ( Site 1002), Boston, Massachusetts
  - University of Michigan ( Site 1006), Ann Arbor, Michigan
  - Vanderbilt University Medical Center-Vanderbilt-Ingram Cancer Center ( Site 1005), Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center-Genitourinary Medical Oncology ( Site 1007), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/